CLINICAL TRIAL: NCT01607944
Title: The Extrapancreatic Metabolic Effects of Incretin Hormones
Brief Title: Incretins and Metabolism
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Associate Professor, Rigshospitalet, Denmark
Other Study IDs: NNF2012
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Glucose Tolerance
- Type 2 Diabetes

SUMMARY:
Incretin hormones (GLP-1 and GIP) have insulin secretory effects on the pancreas that are glucose dependent. Extrapancreatic effects of incretin hormones are reported, however the glucose dependency of these effects have not been examined. In type 2 diabetes, pancreatic endocrine function and incretin metabolism are impaired. The investigators hypothesize that extrapancreatic effects of incretin hormones are glucose depedent and dysregulated in subjects with type 2 diabetes.

Healthy control subjects and type 2 diabetics will undergo pancreatic clamps. In brief, somatostatin will be infused to inhibit pancreatic endocrine function and basal levels of insulin, glucagon, and growth hormone will be replace via infusion. Metabolic flux will be studied during euglycemic and hyperglycemic stages of the pancreatic clamp. Each subject will undergo 3 trials involving the co-infusion of either saline(Control Trial), GLP-1, or GIP. Glucose metabolism will be assessed using 13C-glucose stable isotope methodology combined with indirect calorimetry and expired breath isotope ratio analysis. Blood flow and flow-mediated dilation will be measured using ultrasound Doppler. Skeletal muscle and abdominal adipose biopsies will be taken to examine intracellular signalling.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* BMI 18-35 kg/m2
* NGT or T2DM as classified by ADA criteria

Exclusion Criteria:

* Insulin dependency
* Smokers
* History of or presentation with cardiovascular disease, cancer, and chronic hematological, renal, hepatic, pulmonary disease
* Weight loss (>2 kg in previous 6 months)
* Physical activity (>150 mins/week)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Local community volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Glucose turnover | 0, 1, 2, 3, 4 hours
  Rates of appearance and disappearance (g/min) will be measured by examining [6,6-2H2]glucose enrichment in plasma.

SECONDARY OUTCOMES:
Blood flow and flow-mediated dilation | 0, 1, 2, 3, 4 hours
Palmitate turnover and oxidation | 0, 1, 2, 3, 4 hours
  Rates of appearance and disappearance (g/min) will be measured by examining [U13C]palmitate enrichment in plasma. Rate of oxidation (g/min) will also be measured by examining 13C incorporation into CO2 in expired breath.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Solomon, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark